CLINICAL TRIAL: NCT01027247
Title: OculusGen™ Collagen Matrix Implant for Phaco-Trabeculectomy in Primary Glaucoma: a Case-Control Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Singapore National Eye Centre (Other Government)
Other Study IDs: R539/27/2007
Record Dates: First submitted 2009-12-04; First posted 2009-12-07 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Glaucoma
Keywords: Primary Glaucoma
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Ologen TM

SUMMARY:
Frequently glaucoma is not controlled with clinical treatment ("eyedrops") or laser surgery to control your eye pressure. If this raised pressure is sustained over a long period of time it can lead to permanent damage to the optic nerve (glaucoma) and in severe cases it can result in blindness. You also have cataracts, an opacification of the natural lens inside the eye that is impairing your vision. To prevent further vision loss due to glaucoma, your doctor has recommended glaucoma filtration surgery to lower your eye pressure, and cataract surgery at the same time to improve your sight.

The use of the anti-metabolite (Mitomycin-C) during the operation is currently the drug of choice to improve surgical outcome for glaucoma filtration surgery. Mitomycin-C is a potent antiscarring agent that reduces the amount of scar tissue produced after surgery which leads to better control of eye pressure. Although this potent drug is effective in increasing surgical success, its use is related to a higher risk of post surgical complications, some of which are sight threatening.

The Collagen Matrix Implant is a biodegradable implant (absorbed naturally by tissue), made from porcine collagen, which reduces scar tissue formed after glaucoma filtration surgery without the use of Mitomycin-C. This means that you could be less likely to have a failed glaucoma filtration surgery, and consequently, a poor eye pressure control. In addition, the risk of surgical failure may be reduced because with this technique, we will not be using potent drugs. However, the long-term effect of the OculusGenTm implant in glaucoma filtration surgery is not fully known.

The aim of the study is to determine whether the OculusGenTm implant can equal the success rate of Mitomycin-C in controlling eye pressure, without the potentially sight threatening complications associated with Mitomycin use. And at the same time, this study aim to determine if the implant can reduce potential complications related to glaucoma surgery when compared to the combined surgery augmented with anti-proliferative agents.

This study will recruit 66 subjects from patients attending the Singapore National Eye Centre over a period of 12-24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with primary glaucoma.
2. Age 21 years or over.
3. Uncontrolled glaucoma, with failed medical and laser treatment, requiring trabeculectomy.
4. Visually impairing cataract, requiring cataract extraction surgery.
5. Subject able and willing to cooperate with investigation plan.
6. Subject able and willing to complete postoperative follow-up requirements.
7. Subject willing to sign informed consent form.

Exclusion Criteria:

1. Known allergic reaction to porcine collagen.
2. Vertical cup-disc ratio ≥ 0.9.
3. Patients with secondary glaucoma.
4. Previous intraocular surgery
5. Subject is on warfarin and discontinuation is not recommended.
6. Participation in an investigational study during the 30 days preceding trabeculectomy.
7. Ocular infection within 14 days prior to trabeculectomy.
8. Pregnant or breast-feeding women

   -

Ages: 21 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
To assess the safety and effectiveness of the OculusGenTM Biodegradable Collagen Matrix Implant in Phaco-Trabeculectomy surgeries in patients with Primary Glaucoma